CLINICAL TRIAL: NCT03407742
Title: Strengthening Hispanic Families Via NIDA Prevention Science
Brief Title: Strengthening Hispanic Families Via NIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Principal Investigator, Jose R Parra-Cardona, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1K01DA036747 (NIH)
Record Dates: First submitted 2017-12-01; First posted 2018-01-23 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Adolescent Behavior; Parenting
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of two conditions: (a) intervention consisting of parenting program, or (b) wait-list control group
Who Masked: Participant
Masking Description: Data manager was in charge of conducting randomization and allocating parents to treatment conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): CAPAS Youth Parenting Intervention
  Interventions: Behavioral: CAPAS Youth
- Wait-list control (No Intervention): Participants allocated to this condition were offered the parenting intervention until all T2 assessments of the intervention arm were completed

INTERVENTIONS:
Behavioral: CAPAS Youth — 9-week parenting intervention
  Arms: Intervention

SUMMARY:
The proposed specific aims of this K01 pilot study were:

1. Develop a culturally adapted and web-enhanced version of the Parent Management Training-the Oregon model (GenerationPMTO) intervention for first generation Hispanic families with youth.
2. Implement a small randomized controlled trial (RCT) with the culturally adapted and web-enhanced version of the GenerationPMTO intervention.
3. Systematically examine the implementation feasibility (i.e., rates of engagement, retention, and cultural acceptability) and initial efficacy of the adapted intervention (i.e., reduced parental stress and depression, increased quality of parenting skills, reduced levels of internalizing and externalizing behaviors in youth, and reduced adolescent substance use likelihood).

DETAILED DESCRIPTION:
Recruitment. Participants were recruited according to eligibility criteria, in close collaboration with community partners. Specifically, health and mental health care centers, as well as community organizations and churches were targeted for recruitment activities. Recruitment also consisted of snowball recruitment from participants exposed to the intervention.

General Description of the Intervention. The Parent Management Training-Oregon model (GenerationPMTO) intervention is delivered primarily to parents in order to strengthen parenting skills in a safe learning environment that empower parents to implement these skills at home. The development of the original GenerationPMTO Spanish manual was conducted by Dr. Domenech-Rodriguez according to a comprehensive model of cultural adaptation research.

The intervention consisted of GenerationPMTO and culturally-focused sessions. The GenerationPMTO-focused sessions are detailed in the core treatment manual and have been translated into Spanish utilizing a rigorous process of translation and consultation with Hispanic scholars. Culturally-focused sessions integrated content from three sources. First, we informed sessions according to relevant literature focused on biculturalism. We also informed the intervention by addressing specific cultural themes that were identified as salient in our qualitative studies, which correspond to existing literature on risk and protective factors associated with Hispanic youth. Finally, parents were invited to reflect on additional cultural values and experiences that they consider relevant to their parenting efforts.

With regard to content of individual sessions, module 1 addressed issues associated with immigration, Hispanic culture, and bicultural frameworks. Module 2 addressed issues associated with parenting and biculturalism. Modules 3-6 covered the GenerationPMTO core components as they apply to adolescent populations. Module 7 consists of an in-person session to refine and troubleshoot parenting skills that parents may consider particularly challenging. To enhance the cultural relevance of GenerationPMTO components, we will present all GenerationPMTO parenting skills according to bicultural frameworks, a strategy highly effective the R34 study.

Modules 8-9 reinforced issues of biculturalism having exposed parents to all PMTO core components. A strong focus on biculturalism is particularly relevant as empirical research has demonstrated that the promotion of biculturalism constitutes an effective protective factor for Hispanic youth in first generation Hispanic families.

Randomization. The individual family was the unit of computer-derived randomization, with PTMO-control balance sought for (a) gender of target youth, and (b) time of recruitment. Assessments. Data collection was completed after recruitment (T1) and upon intervention completion (T2).

Intervention Delivery. The intervention was delivered in a major faith-based organization as this site was the preferred site selected by Latino/a parents. In addition to the parenting intervention, a strong advocacy approach was implemented to address various needs of parents (e.g., referral to job training programs or immigration services).

Analyses. Tests of the primary hypothesis will involve fitting of the more assumption-laden subject-specific multivariate response model to Likelihood of Youth Substance Use (LYUS) sub-scale values, followed by fitting of the somewhat more conservative Generalized Estimating Equations (GEE) marginal model with the advantage of fewer assumptions.Our papers will report crude and covariate-adjusted efficacy estimates from both models, allowing readers to draw inferences based on either or both approaches. These same models are used to test the secondary efficacy hypotheses about program impact on parenting skill levels, youth internalizing/externalizing behaviors, and parent stress levels.

ELIGIBILITY:
Parent Inclusion Criteria:

* 18 years or older.
* Living in a one or two-parent family household.
* At least one parent self-identifies as foreign-born and first generation Hispanic/a immigrant, with one or more US-born 12-14 year old children in middle school.
* Spanish speaking.
* Provide written consent to participate in a parenting intervention trial.
* Have access to phone service in home and have home-based internet access.
* Report a combined annual family income is equal or lower than federal income guidelines for families eligible to receive federal welfare assistance.

Youth inclusion criteria:

* Age 12-14 years old.
* Attending middle school.
* Self-identified as Hispanic or Latino.
* English-, or Spanish-speaking, or bilingual.
* Parent report at least one externalizing problem behavior.

Parent Exclusion Criteria:

* Child Protective Services involvement due to confirmed child abuse or neglect
* History of diagnosis with any severe psychiatric disorder.

Focal Youth exclusion criteria:

* Hispanic validated version of Bird et al. screening test at 'high' level of problem behaviors.
* One or more of the DSM-IV-TR conduct or oppositional defiant or substance use disorders
* Documented sexual abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Parenting Positive Involvement | Measured 4-5 months after T1 measurements
  Measures quality of parenting practices aimed at improving parent-youth relationship. Scale 0-4, with lower scores indicating worse outcome.
Parenting Skills Encouragement | Measured 4-5 months after T1 measurements
  Measures quality of parenting practices aimed at motivating children's self-sufficient behaviors. Scale 0-4 with lower scores indicating worse outcomes.
Parenting Discipline | Measured 4-5 months after T1 measurements
  Measures quality of parental limit setting skills. Scale 0-4 with lower score indicating worse outcome.
Parenting Supervision. | Measured 4-5 months after T1 measurements
  Measures quality of parenting practices focused on monitoring and supervision. Scale 0-4 with lower score indicating worse outcome.
Parenting Family Problem Solving | Measured 4-5 months after T1 measurements
  Measures quality of parenting practices aimed at helping youth develop problem solving skills. Scale 0-4 with lower score indicating worse outcome.
Adolescents' Perceived Risk of Drug Use | Measured 4-5 months after T1 measurements
  Measures changes in youth's perception of drug use. Scale 0-4 with higher score indicating best outcome.
Adolescents' Likelihood of Drug Use. | Measured 4-5 months after T1 measurements
  Measures likelihood of youth engaging in drug use. Scale 0-5 with higher score indicating best outcome. Scale 1-5 with higher score indicating worse outcome.
Revised Behavioral Problem checklist | Measured 4-5 months after T1 measurements
  Measures youth's internalizing and externalizing problematic behaviors. Scale 0-2 with lower scores indicating worse outcomes.

SECONDARY OUTCOMES:
Bicultural Involvement Questionnaire | Measured 4-5 months after T1 measurements
  Measures level of acculturation in parents and youth. Scale 1-5. Lower scores indicate US oriented identity and high score indicate Latino-oriented identity.
Hispanic Stress Inventory | Measure 4-5 months after T1 measurements
  Measurements parental stress characteristic of Hispanic immigrant populations. Score 0-5 with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Parra-Cardona, Ph.D., Principal Investigator — the University of Texas at Austin
Locations (1):
- Steve Hicks School of Social Work, the University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
According to IRB regulations, no identifiable data will be shared, only aggregate data. However, the timing for sharing is not yet determined.